CLINICAL TRIAL: NCT06365359
Title: Systemic Lupus Erythematosus and Chlordecone Impregnation in Martinique
Acronym: LUNEK
Status: Recruiting | Type: Observational
Sponsor: University Hospital Center of Martinique (Other)
Collaborators: Institut Pasteur de Guadeloupe (Unknown); Centre de Ressources Biologiques de la Martinique (CeRBiM) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 23_RIPH2-12
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2025-03-31 (Actual); Status verified 2025-03

CONDITIONS: Systemic Lupus Erythematosus; Renal Disease
Keywords: Systemic Lupus Erythematosus; Chlordecone impregnation; Organochlorine pesticide (chlordecone, p,p'-DDE, βHCH, γHCH, PCB 153); Renal Disease
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Kidney Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood cell collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Lupus patients who consult the Martinique University Hospital
  Interventions: Other: Blood sample for analysis of plasma of organochlorine pesticides concentration; Other: Blood sample for cell collection

INTERVENTIONS:
Other: Blood sample for analysis of plasma of organochlorine pesticides concentration — A 20 mL blood sample will be taken up to 6 months after inclusion of the patient for the analysis of chlordecone and the following organochlorine compounds: p,p'-DDE, βHCH, γHCH, PCB 153. This analysis will be carried out at the Institut Pasteur of Guadeloupe (IPG).
Other: Blood sample for cell collection — A 20 mL blood sample will be taken up to 6 months after inclusion of the patient for the cell collection which will be kept at the CeRBiM.
  This collection will be used for subsequent studies on the immunotoxicity of chlordecone, by studying the cytokine, apoptotic and autoreactive functions of PBMC (Peripheral Blood Mononuclear Cells).

SUMMARY:
Chlordecone, an organochlorine pesticide, was widely used on banana farms in the French West Indies. Studies by Inserm and health authorities have confirmed the contamination of the food chain and the majority of the population of the French West Indies by chlordecone.

Epidemiological studies conducted in the French West Indies have shown that exposure to chlordecone at the levels observed is associated with an increased risk of developing several diseases, including premature birth and prostate cancer. Many of the adverse effects associated with chlordecone could be explained by its estrogenic hormonal properties, and systemic lupus erythematosus (SLE) is an autoimmune disease whose sensitivity to estrogen is well known and is reflected by 1) its clear predominance in women, 2) its predominance in women of childbearing age, 3) its risk of exacerbation in the event of pregnancy.

Chlordecone has the potential to modify the activity of SLE through mechanisms other than its pro-estrogenic effects. In rats, chlordecone was observed to induce alterations such as a reduction in lymphocyte count, thymic atrophy, and a decrease in splenic germinal centers and NK cells.

In a mouse model of systemic lupus erythematosus (SLE), exposure to chlordecone results in increased production of immune complexes and anti-DNA antibodies, which are markers of disease activity and monitoring.

Chlordecone also has a cellular effect that reduces the apoptosis of potentially auto-reactive lymphocytes and stimulates the production of GM-CSF, IL-2, TNF-alpha, and IFN-gamma. The latter is central to the pathophysiology of SLE. While experimental studies suggest a potential impact of chlordecone on SLE, no human studies have been conducted to date, and the chlordecone impregnation of lupus patients in Martinique remains unknown.

The most serious and feared complication of SLE is kidney damage. Kidney damage from the disease and the necessary immunosuppressive treatments can lead to significant morbidity and mortality, including death and end-stage chronic renal failure. Therefore, it is important to manage the disease carefully. Suspected lupus nephritis is confirmed by a renal biopsy, which allows for formal diagnosis and categorization into several classes. Suspected cases are identified by a proteinuria to creatininuria ratio greater than 0.5 g/g (or 24-hour proteinuria greater than 0.5g).

The objective of this project is to determine whether there is a positive association between lupus nephritis occurrence in patients followed by the internal medicine department of the Martinique University Hospital and organochlorine pesticide chlordecone impregnation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with systemic lupus erythematosus according to the ACR 1997 or ACR/EULAR 2019 criteria,
* Present in the active line of the internal medicine department of the Martinique University Hospital since 2005,
* Whose illness has been progressing for at least 3 years,
* Living in Martinique or Guadeloupe for at least 1 year,
* Patients who have given their free, informed and written consent.

Exclusion Criteria:

* Patients for whom kidney disease cannot be authenticated or ruled out (refusal, contraindication or impossibility of renal biopsy),
* Patients without social security coverage,
* Current legal protection,
* Patients who have not given their consent to the use of their data,
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with systemic lupus erythematosus according to the ACR 1997 or ACR/EULAR 2019 criteria
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2026-07-02 (Estimated); Study Completion 2026-09-02 (Estimated)

PRIMARY OUTCOMES:
To estimate the risk of presenting a renal complication of lupus disease based on the level of impregnation with chlordecone in the lupus patients seen at the Martinique University Hospital. | 18 months
  Calculation of the Odds ratio (OR) of having lupus kidney disease according to the plasma chlordecone concentration at baseline.
  Patients classified "M+ = Suffering from lupus kidney disease" will be those for whom the diagnosis was suspected based on a proteinuria to creatininuria ratio greater than 0.5 g/g (or 24-hour proteinuria greater than 0.5g) and confirmed by a kidney biopsy which allows the formal diagnosis of lupus kidney damage, but also its categorization into several classes, depending on the cell proliferation observed.
  The biomarker of exposure to chlordecone will, at a minimum, be dichotomized into two classes according to the median value of the distribution of plasma chlordecone concentration (E-/E+).

SECONDARY OUTCOMES:
To compare the activity of lupus according to the level of impregnation with chlordecone. | 18 months
  Average of SELENA-SLEDAI lupus activity score retrospectively assessed from diagnosis to patient inclusion + number of disease flares since the first diagnostic flare.
To compare the after-effects of lupus according to the level of impregnation with chlordecone. | 18 months
  SLICC/SDI lupus after-effects score in the retrospective analysis of the history of the disease.
To describe the distribution of the plasma concentration of chlordecone in lupus patients followed by the internal medicine department of the Martinique University Hospital. | 18 months
  Distribution of plasma chlordecone concentration and of other organochlorine compounds such as: p,p'-DDE, βHCH, γHCH, PCB 153.
To describe the distribution of the plasma concentration of p,p'-DDE in lupus patients followed by the internal medicine department of the Martinique University Hospital. | 18 months
  Distribution of plasma p,p'-DDE concentration
To describe the distribution of the plasma concentration of βHCH in lupus patients followed by the internal medicine department of the Martinique University Hospital. | 18 months
  Distribution of plasma βHCH concentration
To describe the distribution of the plasma concentration of γHCH in lupus patients followed by the internal medicine department of the Martinique University Hospital. | 18 months
  Distribution of plasma γHCH concentration
To describe the distribution of the plasma concentration of PCB 153 in lupus patients followed by the internal medicine department of the Martinique University Hospital. | 18 months
  Distribution of plasma PCB 153 concentration

CONTACTS AND LOCATIONS:
Overall Officials: Benoît SUZON, PhD, Principal Investigator — University Hospital Center of Martinique
Locations (1):
- University Hospital Center of Martinique, Fort-de-France, France